CLINICAL TRIAL: NCT03273569
Title: Preplacental Delivery Intervention for Uterine Conservation Protocol: a Novel Approach for Management of Placenta Accreta
Brief Title: PDIUC Protocol for Placental Accreta
Acronym: PDIUC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, Assistant lecturer, OBGYN department; principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PDIUC001
Record Dates: First submitted 2017-08-05; First posted 2017-09-06 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Placenta Accreta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Intervention Model Description: Women with placenta accreta at the time of Cesarean delivery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women with placenta accreta (Experimental): PDI-UC protocol
  Interventions: Procedure: PDI-UC protocol

INTERVENTIONS:
Procedure: PDI-UC protocol — Preplacental delivery intervention for uterine conservation protocol starts after delivery of the fetus during Cesarean delivery and consists of delayed cord clamping, intramyometrial injection of vasopressin, subdecidual injection of saline, ligation of the uterine arteries, multiple 8 compression sutures, followed by delivery of the placenta, application of pressure and interrupted sutures if needed

SUMMARY:
The aim of this study is to evaluate a novel protocol to conserve the uterus during Cesarean delivery indicated for placenta accreta.

DETAILED DESCRIPTION:
Placenta accreta is a morbid obstetric condition that describes variable non-physiologic invasion of the placenta into the the uterine wall. The incidence of placenta accreta, as a serious cause of postpartum hemorrhage, has substantially increased secondary to increase the rate of Cesarean delivery. Placenta accreta is primarily managed by peripartum hysterectomy prior to delivery of the placenta to avoid uncontrolled bleeding. However, in addition to the surgical risks, hysterectomy is psychologically morbid to many women particularly younger women and women with low parity. Therefore, several conservative options were studied to provide an alternative for hysterectomy in these women. Our study is designated to evaluate a proposed protocol of multi-step interventions to reduce the anticipated amount of bleeding prior to delivery of the placenta.

ELIGIBILITY:
Inclusion Criteria:

* Women with diagnosis of placenta accreta (US or MRI based diagnosis)
* Women who decline hysterectomy
* Pregnancy at 28 weeks of gestation or beyond
* Women who accept to participate in the study

Exclusion Criteria:

* Emergency Cesarean delivery (women with active bleeding)
* Women with cardiac diseases
* Women with coagulopathy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Uterine conservation | Intra-operative (during the time of Cesarean delivery)
  Successive Uterine conservation; no peripartum hysterectomy needed

SECONDARY OUTCOMES:
Primary postpartum hemorrhage | From delivery of the fetus to 1 hour after delivery of the fetus
  Amount of postpartum bleeding > 1000 ml
Severe primary postpartum hemorrhage | From delivery of the fetus to 1 hour after delivery of the fetus
  Amount of postpartum bleeding > 1500 ml
Bladder injury | Intra-operative (during the time of Cesarean delivery)
  Incidental injury of the bladder during delivery of the placenta or control of bleeding
Bowel injury | Intra-operative (during the time of Cesarean delivery)
  Incidental injury of the bladder during delivery of the placenta or control of bleeding
Surgical site infection | Up to 2 weeks after Cesarean delivery
  Cesarean wound infection
Drop in hemoglobin level | Hemoglobin is checked 1 hour prior to Cesarean delivery and again postoperative (24 and 72 hours after Cesarean delivery)
  Change in hemoglobin before and more than 24 hours after delivery

IPD SHARING:
Plan to Share IPD: No